CLINICAL TRIAL: NCT03916120
Title: Single Nucleotide Polymorphisms (SNPs) Associated With Postoperative Analgesic Failure After Single-port Video-Assisted Thoracoscopic Surgery
Brief Title: Single Nucleotide Polymorphisms (SNPs) Associated With Postoperative Analgesic Failure
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-067
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Thoracic Surgery, Video-Assisted; Polymorphism, Single Nucleotide
MeSH Terms: conditions — Pain, Postoperative | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative Analgesic Failure
  Interventions: Genetic: Genetic analysis
- Postoperative Analgesic Success
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — Collect 2ml intravenous blood from patients after anaesthesia.

SUMMARY:
Postoperative pain remains relatively high within 48h for Chinese patients who receive video-assisted thoracoscopic surgery. Different patients experience different pain intensity. This suggests that there may be genetic variants that make some patients susceptible to analgesic failure. Using blood samples from patients, the investigators are going to analyze the relationship between single nucleotide polymorphisms (SNPs) in genes that are known to be involved in analgesic failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 70 and Age ≥18
* Selective operation lung section with video-assisted thoracic surgery (VATS)
* III ≥ American Society of Anesthesiologists classification (ASA classification) ≥I
* Patients informed and agreed to join the study

Exclusion Criteria:

* Abnormal function of liver and kidney
* Allergic- dependence history of alcohol, opioids and Local anesthetics
* No noncompliance
* Mental disease history，language communication disorder，cicatricial diathesis
* Underweight or overweight（BMI<18 or >30)
* Patients not suitable for clinical subjects for other reasons
* Sedatives, analgesics, antiemetic drugs and anti pruritus drugs were used within 24hours before the operation.
* History of previous abnormal anaesthesia
* Women during pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving single-port video-assisted thoracoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic failure | 8 a.m. at the first day after surgery.
  Once patient experience at least one of the following situations:
  1. Bad patients sleep quality
  2. Require extra analgesic drug
  3. Low satisfaction with pain control
  4. Bolus times > 1 per hour

CONTACTS AND LOCATIONS:
Overall Officials: Min Min, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xing X, Bai Y, Sun K, Yan M. Single nucleotide polymorphisms associated with postoperative inadequate analgesia after single-port VATS in Chinese population. BMC Anesthesiol. 2020 Feb 5;20(1):38. doi: 10.1186/s12871-020-0949-6. PMID 32024468